CLINICAL TRIAL: NCT01798498
Title: Open-label Uncontrolled, Multicenter Study for the Evaluation of the Efficacy and Safety of the Dermal Filler Princess® VOLUME in Nasolabial Folds
Brief Title: Study for the Evaluation of the Efficacy and Safety of the Dermal Filler Princess® VOLUME in Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Croma-Pharma GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVN1
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Princess® VOLUME (Experimental): Injection of Princess® VOLUME into the deep dermis or subcutis of both nasolabial folds.
  A touch-up treatment may be performed at Day 14 if correction is not complete after the first injection.
  The injected volumes will be estimated by the investigator and depend on the depth of the nasolabial folds
  Interventions: Device: Princess® VOLUME

INTERVENTIONS:
Device: Princess® VOLUME
  Other Names: highly cross-linked, viscoelastic hyaluronic acid injectable gel implant

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy and safety of Princess® VOLUME for the correction of nasolabial folds.

ELIGIBILITY:
Major Inclusion Criteria:

* Male or female subjects between 30 years and 65 years
* Wrinkle score of at least 2 according to the Modified Fitzpatrick Wrinkle Scale (MFWS)

Major Exclusion Criteria:

* For females: pregnancy, lactating, planned pregnancy or unwilling to use contraceptives
* History of allergic reaction to hyaluronic acid products
* Facial surgery or implantation of dermal fillers in the nasolabial region within the last 24 months
* Skin of the nasolabial region affected by cosmetic treatments (e.g. laser therapy within the last 12 months, chemical peeling within the last 3 months, dermabrasion within the last 12 months, botulinum toxin within the last 12 months )
* Connective tissue diseases
* Diabetes mellitus or uncontrolled systemic diseases
* Known human immune deficiency virus-positive individuals
* Presence of silicone implant or another non-absorbable substance (permanent fillers) in the area of product application
* Cutaneous lesions in the evaluated area
* Tendency to keloid formation and/or hypertrophic scars
* Autoimmune disease
* History of allergies against cosmetic filling products and re-current herpes simplex
* History of immune system degradation

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Kopera, Prof. Dr., Principal Investigator — Department of Dermatology and Gerontology, Medical University Graz
Locations (3):
- Austria (3):
  - Medical University Graz, Graz
  - Ordination 1, Vienna
  - Ordination 2, Vienna

RESULTS

PARTICIPANT FLOW:
Groups:
- Princess® VOLUME: Subjects received one injection of the investigational device to both nasolabial folds on Day 0. After the initial treatment, a touch-up treatment was permitted on Day 14, if full correction of the wrinkle had not been achieved with the baseline treatment.
  The volume of application depended on the depth of wrinkle to be corrected and was chosen by the investigator.
Period: Overall Study
Arm/Group | Princess® VOLUME
Started | 48
Completed | 47
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 1 Subject was lost to follow up after Day 14
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 52 [31 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Fitzpatrick Wrinkle Scale (MFWS) From Day 0 to Day 180
Description: The primary efficacy endpoint was the absolute change in MFWS from Day 0 to Day 180
  The Modified Fitzpatrick Wrinkle Scale (MFWS), an established objective and validated measurement for nasolabial wrinkle severity assessments.
  The MFWS is a 7-point rating scale ranging from 0 = no wrinkle to 3 = deep wrinkle where grades are defined as follow:
  Grade Definition 0 No wrinkle: no visible wrinkle, continuous skin line 0.5 Very shallow yet visible wrinkle
  1. Fine wrinkle: visible wrinkle and slight indentation 1.5 Visible wrinkle and clear indentation, <1 mm wrinkle depth
  2. Moderate wrinkle: clear visible wrinkle 1 - 2 mm wrinkle 2.5 Prominent and visible wrinkle: more than 2 mm and less than 3 mm wrinkle depth
  3. Deep wrinkle: deep and furrow wrinkle; more than 3 mm wrinkle depth
Time Frame: From Day 0 to Day 180
Population: safety analysis set (SAF) - The SAF included all subjects who received the investigational device at least once.
  The mean of both measurements (right/left nasolabial fold) is used.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 47
score on a scale | -1.309 (0.373)

2. Secondary Outcome: Change in the Modified Fitzpatrick Wrinkle Scale (MFWS) From Day 0 to Days 30, 90, and 270
Description: The change in absolute Modified Fitzpatrick Wrinkle Scale (MFWS) from Day 0 was additionally assessed at Days 30, 90, and 270
  The Modified Fitzpatrick Wrinkle Scale (MFWS), an established objective and validated measurement for nasolabial wrinkle severity assessments
  The MFWS is a 7-point rating scale ranging from 0 = no wrinkle to 3 = deep wrinkle where grades are defined as follow:
  Grade Definition 0 No wrinkle: no visible wrinkle, continuous skin line 0.5 Very shallow yet visible wrinkle
  1. Fine wrinkle: visible wrinkle and slight indentation 1.5 Visible wrinkle and clear indentation, <1 mm wrinkle depth
  2. Moderate wrinkle: clear visible wrinkle 1 - 2 mm wrinkle 2.5 Prominent and visible wrinkle: more than 2 mm and less than 3 mm wrinkle depth
  3. Deep wrinkle: deep and furrow wrinkle; more than 3 mm wrinkle depth
Time Frame: Day 0 to Days 30, 90, and 270
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 47
score on a scale
  change in MFWS at Day 30 | -1.484 (0.408)
  change in MFWS at Day 90 | -1.436 (0.415)
  change in MFWS at Day 270 | -1.223 (0.401)

3. Secondary Outcome: Percentage of Subjects With an Improvement of at Least 0.5 on the Modified Fitzpatrick Wrinkle Scale (MFWS)
Description: Percentage of subjects with an improvement of at least 0.5 on the Modified Fitzpatrick Wrinkle Scale (MFWS) at Days 30, 90, 180, and 270
  The Modified Fitzpatrick Wrinkle Scale (MFWS), an established objective and validated measurement for nasolabial wrinkle severity assessments
  The MFWS is a 7-point rating scale ranging from 0 = no wrinkle to 3 = deep wrinkle where grades are defined as follow:
  Grade Definition 0 No wrinkle: no visible wrinkle, continuous skin line 0.5 Very shallow yet visible wrinkle
  1. Fine wrinkle: visible wrinkle and slight indentation 1.5 Visible wrinkle and clear indentation, <1 mm wrinkle depth
  2. Moderate wrinkle: clear visible wrinkle 1 - 2 mm wrinkle 2.5 Prominent and visible wrinkle: more than 2 mm and less than 3 mm wrinkle depth
  3. Deep wrinkle: deep and furrow wrinkle; more than 3 mm wrinkle depth
Time Frame: Days 30, 90, 180, and 270
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 47
Participants
  Improvement of at least 0.5 Scores on the MFWS - day 30 | 47
  Improvement of at least 0.5 Scores on the MFWS - day 90 | 47
  Improvement of at least 0.5 Scores on the MFWS - day 180 | 47
  Improvement of at least 0.5 Scores on the MFWS - day 270 | 47

4. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction at Days 30, 90, 180, and 270
  To assess subject's satisfaction, subjects were asked to indicate their level of satisfaction on 3- or 5-point scales as follows:
  * Question 1: How would you judge the change of your appearance after treatment (asked at Days 30, 90, 180, and 270):
    1. Very much improved
    2. Much improved
    3. Slightly improved
    4. No change
    5. Worsened
  * Question 2: How satisfied are you with the treatment (to be asked at Days 30 and 270):
    1. Very satisfied
    2. Satisfied
    3. Not satisfied
  * Question 3: Would you recommend the treatment to your friends and acquaintances (to be asked at Days 30 and 270):
    1. Yes
    2. Perhaps
    3. No
Time Frame: Days 30, 90, 180, and 270
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 47
Participants
  Day 30 : Q1 - Appearance after treatment - very much improved | 16
  Day 30 : Q1 - Appearance after treatment - much improved | 27
  Day 30 : Q1 - Appearance after treatment - sligthly improved | 4
  Day 30 : Q1 - Appearance after treatment - no change | 0
  Day 30 : Q1 - Appearance after treatment - worsened | 0
  Day 30 : Q2 - Satisfaction with treatment - very satisfied | 42
  Day 30 : Q2 - Satisfaction with treatment - satisfied | 5
  Day 30 : Q2 - Satisfaction with treatment - not satisfied | 0
  Day 30 : Q3 - Recommendation of treatment - yes | 46
  Day 30 : Q3 - Recommendation of treatment - perhaps | 1
  Day 30 : Q3 - Recommendation of treatment - no | 0
  Day 90 : Q1 - Appearance after treatment - very much improved | 6
  Day 90 : Q1 - Appearance after treatment - much improved | 37
  Day 90 : Q1 - Appearance after treatment - sligthly improved | 4
  Day 90 : Q1 - Appearance after treatment - no change | 0
  Day 90 : Q1 - Appearance after treatment - worsened | 0
  Day 90 : Q2 - Satisfaction with treatment - very satisfied: number analyzed (Participants) | 0
  Day 90 : Q2 - Satisfaction with treatment - satisfied: number analyzed (Participants) | 0
  Day 90 : Q2 - Satisfaction with treatment - not satisfied: number analyzed (Participants) | 0
  Day 90 : Q3 - Recommendation of treatment - yes: number analyzed (Participants) | 0
  Day 90 : Q3 - Recommendation of treatment - perhaps: number analyzed (Participants) | 0
  Day 90 : Q3 - Recommendation of treatment - no: number analyzed (Participants) | 0
  Day 180 : Q1 - Appearance after treatment - very much improved | 2
  Day 180 : Q1 - Appearance after treatment - much improved | 30
  Day 180 : Q1 - Appearance after treatment - sligthly improved | 15
  Day 180 : Q1 - Appearance after treatment - no change | 0
  Day 180 : Q1 - Appearance after treatment - worsened | 0
  Day 180 : Q2 - Satisfaction with treatment - very satisfied: number analyzed (Participants) | 0
  Day 180 : Q2 - Satisfaction with treatment - satisfied: number analyzed (Participants) | 0
  Day 180 : Q2 - Satisfaction with treatment - not satisfied: number analyzed (Participants) | 0
  Day 180 : Q3 - Recommendation of treatment - yes: number analyzed (Participants) | 0
  Day 180 : Q3 - Recommendation of treatment - perhaps: number analyzed (Participants) | 0
  Day 180 : Q3 - Recommendation of treatment - no: number analyzed (Participants) | 0
  Day 270 : Q1 - Appearance after treatment - very much improved | 5
  Day 270 : Q1 - Appearance after treatment - much improved | 25
  Day 270 : Q1 - Appearance after treatment - sligthly improved | 15
  Day 270 : Q1 - Appearance after treatment - no change | 2
  Day 270 : Q1 - Appearance after treatment - worsened | 0
  Day 270 : Q2 - Satisfaction with treatment - very satisfied | 38
  Day 270 : Q2 - Satisfaction with treatment - satisfied | 8
  Day 270 : Q2 - Satisfaction with treatment - not satisfied | 1
  Day 270 : Q3 - Recommendation of treatment - yes | 44
  Day 270 : Q3 - Recommendation of treatment - perhaps | 3
  Day 270 : Q3 - Recommendation of treatment - no | 0

5. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS)
Description: Investigator rating of aesthetic improvement based on GAIS
  The GAIS is a 5-point scale that rates global aesthetic improvement in appearance, compared to pre-treatment, as judged by the investigator. The rating categories were 'worse', 'no change', 'improved', 'much improved', and 'very much improved'.
Time Frame: Days 14, 30, 90, 180, 270
Population: safety analysis set (SAF) - The SAF included all subjects who received the investigational device at least once.The mean of both measurements (right/left nasolabial fold) is used.
Measure: Count of Participants; unit: Participants
Groups:
- Princess® VOLUME: Subjects received one injection of the investigational device to both nasolabial folds (NLFs) on Day 0. After the initial treatment, a touch-up treatment was permitted on Day 14, if full correction of the wrinkle had not been achieved with the baseline treatment.
  The volume of application depended on the depth of wrinkle to be corrected and was chosen by the investigator.
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 48
Participants
  Day 14 - right NLF: very much improved | 14
  Day 14 - right NLF: much improved | 29
  Day 14 - right NLF: improved | 5
  Day 14 - right NLF: no change | 0
  Day 14 - right NLF: worse | 0
  Day 14 - left NLF: very much improved | 13
  Day 14 - left NLF: much improved | 27
  Day 14 - left NLF: improved | 8
  Day 14 - left NLF: no change | 0
  Day 14 - left NLF: worse | 0
  Day 30 - right NLF: number analyzed (Participants) | 47
  Day 30 - right NLF: very much improved | 14
  Day 30 - right NLF: much improved | 32
  Day 30 - right NLF: improved | 1
  Day 30 - right NLF: no change | 0
  Day 30 - right NLF: worse | 0
  Day 30 - left NLF: number analyzed (Participants) | 47
  Day 30 - left NLF: very much improved | 15
  Day 30 - left NLF: much improved | 30
  Day 30 - left NLF: improved | 2
  Day 30 - left NLF: no change | 0
  Day 30 - left NLF: worse | 0
  Day 90 - right NLF: number analyzed (Participants) | 47
  Day 90 - right NLF: very much improved | 11
  Day 90 - right NLF: much improved | 35
  Day 90 - right NLF: improved | 1
  Day 90 - right NLF: no change | 0
  Day 90 - right NLF: worse | 0
  Day 90 - left NLF: number analyzed (Participants) | 47
  Day 90 - left NLF: very much improved | 11
  Day 90 - left NLF: much improved | 33
  Day 90 - left NLF: improved | 3
  Day 90 - left NLF: no change | 0
  Day 90 - left NLF: worse | 0
  Day 180 - right NLF: number analyzed (Participants) | 47
  Day 180 - right NLF: very much improved | 5
  Day 180 - right NLF: much improved | 36
  Day 180 - right NLF: improved | 6
  Day 180 - right NLF: no change | 0
  Day 180 - right NLF: worse | 0
  Day 180 - left NLF: number analyzed (Participants) | 47
  Day 180 - left NLF: very much improved | 5
  Day 180 - left NLF: much improved | 32
  Day 180 - left NLF: improved | 9
  Day 180 - left NLF: no change | 1
  Day 180 - left NLF: worse | 0
  Day 270 - right NLF: number analyzed (Participants) | 47
  Day 270 - right NLF: very much improved | 4
  Day 270 - right NLF: much improved | 33
  Day 270 - right NLF: improved | 9
  Day 270 - right NLF: no change | 1
  Day 270 - right NLF: worse | 0
  Day 270 - left NLF: number analyzed (Participants) | 47
  Day 270 - left NLF: very much improved | 4
  Day 270 - left NLF: much improved | 31
  Day 270 - left NLF: improved | 11
  Day 270 - left NLF: no change | 1
  Day 270 - left NLF: worse | 0

6. Other Pre Specified Outcome: Modified Fitzpatrick Wrinkle Scale (MFWS) Grades Per Day
Description: Percentage of subjects with an improvement of at least 0.5 on the Modified Fitzpatrick Wrinkle Scale (MFWS) at Days 14, 30, 90, 180, and 270
  The Modified Fitzpatrick Wrinkle Scale (MFWS), an established objective and validated measurement for nasolabial wrinkle severity assessments
  The MFWS is a 7-point rating scale ranging from 0 = no wrinkle to 3 = deep wrinkle where grades are defined as follow:
  Grade Definition 0 No wrinkle: no visible wrinkle, continuous skin line 0.5 Very shallow yet visible wrinkle
  1. Fine wrinkle: visible wrinkle and slight indentation 1.5 Visible wrinkle and clear indentation, <1 mm wrinkle depth
  2. Moderate wrinkle: clear visible wrinkle 1 - 2 mm wrinkle 2.5 Prominent and visible wrinkle: more than 2 mm and less than 3 mm wrinkle depth
  3. Deep wrinkle: deep and furrow wrinkle; more than 3 mm wrinkle depth
Time Frame: Day 0 to Day 14, 30, 90, 180, and 270
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 48
Participants
  Day 0 - right NLF: Grade 0 | 0
  Day 0 - right NLF: Grade 0.5 | 0
  Day 0 - right NLF: Grade 1 | 0
  Day 0 - right NLF: Grade 1.5 | 0
  Day 0 - right NLF: Grade 2 | 30
  Day 0 - right NLF: Grade 2.5 | 16
  Day 0 - right NLF: Grade 3 | 2
  Day 0 - left NLF: Grade 0 | 0
  Day 0 - left NLF: Grade 0.5 | 0
  Day 0 - left NLF: Grade 1 | 0
  Day 0 - left NLF: Grade 1.5 | 0
  Day 0 - left NLF: Grade 2 | 26
  Day 0 - left NLF: Grade 2.5 | 19
  Day 0 - left NLF: Grade 3 | 3
  Day 14 - right NLF: Grade 0 | 4
  Day 14 - right NLF: Grade 0.5 | 18
  Day 14 - right NLF: Grade 1 | 19
  Day 14 - right NLF: Grade 1.5 | 7
  Day 14 - right NLF: Grade 2 | 0
  Day 14 - right NLF: Grade 2.5 | 0
  Day 14 - right NLF: Grade 3 | 0
  Day 14 - left NLF: Grade 0 | 6
  Day 14 - left NLF: Grade 0.5 | 11
  Day 14 - left NLF: Grade 1 | 24
  Day 14 - left NLF: Grade 1.5 | 7
  Day 14 - left NLF: Grade 2 | 0
  Day 14 - left NLF: Grade 2.5 | 0
  Day 14 - left NLF: Grade 3 | 0
  Day 30 - right NLF: number analyzed (Participants) | 47
  Day 30 - right NLF: Grade 0 | 4
  Day 30 - right NLF: Grade 0.5 | 18
  Day 30 - right NLF: Grade 1 | 22
  Day 30 - right NLF: Grade 1.5 | 3
  Day 30 - right NLF: Grade 2 | 0
  Day 30 - right NLF: Grade 2.5 | 0
  Day 30 - right NLF: Grade 3 | 0
  Day 30 - left NLF: number analyzed (Participants) | 47
  Day 30 - left NLF: Grade 0 | 5
  Day 30 - left NLF: Grade 0.5 | 16
  Day 30 - left NLF: Grade 1 | 24
  Day 30 - left NLF: Grade 1.5 | 2
  Day 30 - left NLF: Grade 2 | 0
  Day 30 - left NLF: Grade 2.5 | 0
  Day 30 - left NLF: Grade 3 | 0
  Day 90 - right NLF: number analyzed (Participants) | 47
  Day 90 - right NLF: Grade 0 | 4
  Day 90 - right NLF: Grade 0.5 | 15
  Day 90 - right NLF: Grade 1 | 25
  Day 90 - right NLF: Grade 1.5 | 3
  Day 90 - right NLF: Grade 2 | 0
  Day 90 - right NLF: Grade 2.5 | 0
  Day 90 - right NLF: Grade 3 | 0
  Day 90 - left NLF: number analyzed (Participants) | 47
  Day 90 - left NLF: Grade 0 | 4
  Day 90 - left NLF: Grade 0.5 | 13
  Day 90 - left NLF: Grade 1 | 27
  Day 90 - left NLF: Grade 1.5 | 3
  Day 90 - left NLF: Grade 2 | 0
  Day 90 - left NLF: Grade 2.5 | 0
  Day 90 - left NLF: Grade 3 | 0
  Day 180 - right NLF: number analyzed (Participants) | 47
  Day 180 - right NLF: Grade 0 | 1
  Day 180 - right NLF: Grade 0.5 | 14
  Day 180 - right NLF: Grade 1 | 25
  Day 180 - right NLF: Grade 1.5 | 6
  Day 180 - right NLF: Grade 2 | 1
  Day 180 - right NLF: Grade 2.5 | 0
  Day 180 - right NLF: Grade 3 | 0
  Day 180 - left NLF: number analyzed (Participants) | 47
  Day 180 - left NLF: Grade 0 | 1
  Day 180 - left NLF: Grade 0.5 | 13
  Day 180 - left NLF: Grade 1 | 26
  Day 180 - left NLF: Grade 1.5 | 5
  Day 180 - left NLF: Grade 2 | 2
  Day 180 - left NLF: Grade 2.5 | 0
  Day 180 - left NLF: Grade 3 | 0
  Day 270 - right NLF: number analyzed (Participants) | 47
  Day 270 - right NLF: Grade 0 | 0
  Day 270 - right NLF: Grade 0.5 | 14
  Day 270 - right NLF: Grade 1 | 20
  Day 270 - right NLF: Grade 1.5 | 12
  Day 270 - right NLF: Grade 2 | 0
  Day 270 - right NLF: Grade 2.5 | 0
  Day 270 - right NLF: Grade 3 | 1
  Day 270 - left NLF: number analyzed (Participants) | 47
  Day 270 - left NLF: Grade 0 | 0
  Day 270 - left NLF: Grade 0.5 | 13
  Day 270 - left NLF: Grade 1 | 23
  Day 270 - left NLF: Grade 1.5 | 10
  Day 270 - left NLF: Grade 2 | 0
  Day 270 - left NLF: Grade 2.5 | 1
  Day 270 - left NLF: Grade 3 | 0

7. Other Pre Specified Outcome: Improvement in MFWS in One or Both Nasolabial Folds Over Time
Description: Percentage of subjects with an improvement of at least 0.5 on the Modified Fitzpatrick Wrinkle Scale (MFWS) from Day 0 to Days 30, 90, 180, and 270
  The Modified Fitzpatrick Wrinkle Scale (MFWS), an established objective and validated measurement for nasolabial wrinkle severity assessments.
  The MFWS is a 7-point rating scale ranging from 0 = no wrinkle to 3 = deep wrinkle where grades are defined as follow:
  Grade Definition 0 No wrinkle: no visible wrinkle, continuous skin line 0.5 Very shallow yet visible wrinkle
  1. Fine wrinkle: visible wrinkle and slight indentation 1.5 Visible wrinkle and clear indentation, <1 mm wrinkle depth
  2. Moderate wrinkle: clear visible wrinkle 1 - 2 mm wrinkle 2.5 Prominent and visible wrinkle: more than 2 mm and less than 3 mm wrinkle depth
  3. Deep wrinkle: deep and furrow wrinkle; more than 3 mm wrinkle depth
Time Frame: Day 0 to Day 30, 90, 180, and 270
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Princess® VOLUME
Number analyzed (Participants) | 47
Participants
  Day 30 : 0.5 both NLFs | 47
  Day 30 : 1.0 one NLF | 46
  Day 30 : 1.0 both NLFs | 46
  Day 30 : 1.5 one NLF | 36
  Day 30 : 1.5 both NLFs | 29
  Day 30 : 2.0 one NLF | 15
  Day 30 : 2.0 both NLFs | 10
  Day 90 : 0.5 both NLFs | 47
  Day 90 : 1.0 one NLF | 46
  Day 90 : 1.0 both NLFs | 45
  Day 90 : 1.5 one NLF | 33
  Day 90 : 1.5 both NLFs | 27
  Day 90 : 2.0 one NLF | 14
  Day 90 : 2.0 both NLFs | 9
  Day 180 : 0.5 both NLFs | 47
  Day 180 : 1.0 one NLF | 45
  Day 180 : 1.0 both NLFs | 42
  Day 180 : 1.5 one NLF | 30
  Day 180 : 1.5 both NLFs | 22
  Day 180 : 2.0 one NLF | 10
  Day 180 : 2.0 both NLFs | 3
  Day 270 : 0.5 both NLFs | 46
  Day 270 : 1.0 one NLF | 43
  Day 270 : 1.0 both NLFs | 40
  Day 270 : 1.5 one NLF | 26
  Day 270 : 1.5 both NLFs | 19
  Day 270 : 2.0 one NLF | 7
  Day 270 : 2.0 both NLFs | 2

ADVERSE EVENTS:
Arm/Group | Princess® VOLUME
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 12/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Princess® VOLUME (N=48)
Uterin Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Princess® VOLUME (N=48)
Hematoma (General disorders) | 9 (9)
bruising (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes